CLINICAL TRIAL: NCT02024451
Title: Comparison of the Effect of Radial Shock Wave and Acupuncture in the Treatment of Myofascial Pain Syndrome
Brief Title: Radial Shock Wave and Acupuncture for Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20130712R
Record Dates: First submitted 2013-12-03; First posted 2013-12-31 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Myofascial Pain
Keywords: Radial shock wave; Acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radial shock wave, Acupuncture (Active Comparator): Radial shock wave: 2 Hz with 2000 shock waves, and the energy level of 0.056mJ/mm2 in the trapezius muscle. It will be done once per week for 3 weeks.
  Acupuncture: performed at Fenfchi (GB20) point over upper back. It will be performed once per week for 3 weeks .
  Interventions: Device: Radial shock wave; Device: Acupuncture
- radial shock wave& no treatment (No Intervention): No treatment: patients recieved no intervention.

INTERVENTIONS:
Device: Radial shock wave — radial shock wave: Treatment point is the origin attachment of upper trapezius at the external occipital protuberance. Radial shock wave therapy will be performed once per week, and will be continued for 3 weeks. Acetaminophen will be prescribed as rescue medication, and the amount given will be recorded at the end of the study.
  Other Names: Dolorclast
  Arms: Radial shock wave, Acupuncture
Device: Acupuncture — Acupuncture is performed at Fenfchi (GB20) point over upper back by the same physiatrist to all patients.
  Arms: Radial shock wave, Acupuncture

SUMMARY:
Myofascial pain syndrome is common in Rehabilitation clinic. The pain occurs asymmetrically in isolated or regional muscles, and is associated with acute muscle strain or chronic muscle overuse. Myofascial pain is characteristics with localized muscle tenderness, palpable intramuscular taut band, typical referred pain, and local twitch response.

Treatment of myofascial pain syndrome includes physical therapy, stretch exercise, dry needle insertion and trigger point injection. Acupuncture originated from ancient Chinese medicine which involves the insertion of fine needle to stimulate specific points of the body along the 12 meridians. The mechanism of pain relief may be initiated by activation of both spinal segmental and supraspinal centers. Acupuncture is commonly used for pain relief.

Recently, radial shock wave has been shown to be effective in the treatment of chronic musculoskeletal pain, including calcific tendinitis, epicondylitis, and plantar fasciitis. The energy and pressure produced by radial shock wave is focused on the treated musculoskeletal tissue. The mechanism of action has been hypothesized that the energy could result in analgesic effect and stimulation of angiogenesis and healing response and then relief of the symptoms. The effectiveness of radial shock wave on treatment of myofascial pain was reported by Jeon and colleagues in 2012.

The aim of this study is to compare the efficacy of acupuncture and radial shock wave therapy in patients with myofascial pain syndrome.

DETAILED DESCRIPTION:
80 participants diagnosed with myofascial pain syndrome in trapezius muscle will be enrolled from the outpatient clinic of Department of Physical Medicine and Rehabilitation in Shin Kong Wu Ho-Su Memorial Hospital .

The patients will be randomized to either treatment groups: group 1, radial extracorporeal shock wave therapy (RSWT group) and group 2, acupuncture group (AC group).

All treatments will be given in the Department of Physical Medicine and Rehabilitation, and will be handled by a physiatrist who is familiar with both kinds of therapy.

The RSWT is delivered at 2 Hz with 2000 shock waves and the energy level of 0.056 mJ / mm2 in the trapezius muscle. Treatment point is the origin attachment of upper trapezius at the external occipital protuberance. RSWT will be performed once per week, and will be continued for 3 weeks.

Acupuncture is performed at Fenfchi (GB20) point over upper back. This acupoint is a common local point for treating upper back pain. Acupuncture therapy will be provided by the same physiatrist to all patients.

The primary outcome measures are VAS for pain and pain threshold. The secondary outcome measures are neck disability index, and patients' satisfaction. All subjects will be assessed by an independent, blinded investigator at baseline, post treatment and at 1-month after the treatments are completed.

Demographic data, including age, sex, employment status, and sleep quality, history of head or neck surgery, or other psychiatric and medical disorders will be recorded at baseline. A history will be taken concerning the duration of complaints (months), previous treatments (injections, physical therapy), and current pain medications. Concomitant diseases and the use of medications will be registered.

ELIGIBILITY:
Inclusion Criteria:Physical examination showed

* unilateral upper back pain,
* palpable intramuscular taut band,
* normal neurological examination
* presence of trigger points

Exclusion Criteria:

* bilateral neck pain
* pregnancy
* coagulopathy
* patients with pacemaker
* open wound at treatment area
* cervical spine fracture or previous operation around neck
* cervical myelopathy
* rheumatoid arthritis
* severe systemic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
VAS for pain | up to 1 week before treatment, on the day treatment is completed, 1 month after treatment completed
  horizontal lines of 100 mm, with 0 indicating no pain on the left and 100 indicating very severe pain on the right
Pain threshold | up to 1 week before treatment, on the day treatment is completed, 1 month after treatment completed
  A pressure algometer, the pressure threshold meter, was applied onto the affected and unaffected sides of upper trapezius, with the metal rod perpendicular to the surface of the skin. The pressure of compression was increased gradually until the subject began to feel pain or any discomfort. Three repetitive measurements at an interval of 20-60 s were performed. The average values of the three readings were used for data analysis of the pain threshold measurement.

SECONDARY OUTCOMES:
neck disability index | up to 1 week before treatment, on the day treatment is completed, 1 month after treatment completed
  It consists of 10 items referring to various activities (personal care, lifting, driving, work, sleeping, concentrating, reading, recreation) and pain (pain intensity, headache) with six possible answers for each item, only one answer to be chosen by the patient for each item. Scores for each item ranged from 0 (no pain and functional limitation) to 5 (worst pain and maximal limitation), resulting in a total score of 0 (not disabled) to 50 (totally disabled).
cervical active range of motion | up to 1 week before treatment, on the day treatment is completed, 1 month after treatment completed
  neck flexion, extension, rotation and side bending

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ling Chen, MD, Principal Investigator — Shin Kong Hospital,No. 95, Wen Chang Road, Shih Lin District, Taipei City, Twiwan
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taipei city, Taiwan

REFERENCES:
- [Result] Jeon JH, Jung YJ, Lee JY, Choi JS, Mun JH, Park WY, Seo CH, Jang KU. The effect of extracorporeal shock wave therapy on myofascial pain syndrome. Ann Rehabil Med. 2012 Oct;36(5):665-74. doi: 10.5535/arm.2012.36.5.665. Epub 2012 Oct 31. PMID 23185731